CLINICAL TRIAL: NCT01170143
Title: A Randomized Study to Investigate the Efficacy and Safety of qw or q3w Trastuzumab, Paclitaxel and Carboplatin in Patients With IIB-IIIB HER2 Positive Breast Cancer
Brief Title: Efficacy and Safety Study of Trastuzumab, Paclitaxel and Carboplatin on HER2+ Preoperative Breast Cancer
Acronym: PCH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Zhimin Shao/professor, Cancer Hospital Affiliated to Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22700
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: IIB-IIIB Breast Cancer; Her2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab QW (Active Comparator): Arm A: Trastuzumab 2mg/kg, d1; qw (loading dose 4mg/kg wk1) Paclitaxel 80mg/m2,. d1; qw Carboplatin AUC 2 d1, qw
  Interventions: Drug: Trastuzumab QW, Trastuzumab Q3W
- Trastuzumab Q3W (Active Comparator): Arm B: Trastuzumab 6mg/kg, d1(loading dose 8mg/kg wk1) Paclitaxel 175mg/m2,. d1, q3w; Carboplatin AUC 6 ,. d1,q3w
  Interventions: Drug: Trastuzumab QW, Trastuzumab Q3W

INTERVENTIONS:
Drug: Trastuzumab QW, Trastuzumab Q3W — two arms using Trastuzumab QW vs Q3W
  Other Names: Herceptin

SUMMARY:
To compare the efficacy in terms of the pathological complete response rate (pCR) to preoperative administration of qw or q3w Paclitaxel, Carboplatin and Trastuzumab (PCH)

DETAILED DESCRIPTION:
Currently Herceptin has moved to Neoadjuvant treatment combined with chemotherapy. Paclitaxel and Carboplatin are two of the best partners with high pCR. The significant efficacy and good safety profile of Herceptin® combination with taxane as adjuvant treatment on EBC are accepted; 1 year of Herceptin as adjuvant treatment is one standard therapy. This study is one small Phase II trial to explore the efficacy and safety of QW and Q3W of PCH as Neoadjuvant treatment, we only plan 60 pts and the trend of the two curves is anticipated

ELIGIBILITY:
Inclusion Criteria:

1. Women aged equals to or more than 18 years and no more than 70 years with life expectancy more than 12 months
2. Histologically confirmed invasive breast cancer (excluding inflammatory breast cancer) by core needle biopsy, T2N1 or local advanced breast cancer, with no evidence of metastasis
3. HER2 positive confirmed by FISH/CISH+ or IHC 3+
4. With no history of cancer other than in situ uterine cervix cancer or skin basal cell carcinoma
5. Adequate hematopoietic function: Neutrophil larger than 1.5*109/L; Hb larger than 100g/L; PLT larger than 100*109/L
6. Adequate hepatic and renal function

   * serum AST less than 60U/L
   * Total bilirubin less than 1.5 ULN
   * serum creatinine less than 110umol/L
   * BUN less than 7.1mmol/L
7. LVEF 55% by MUGA scan or echocardiography
8. Adequate coagulation function
9. ECOG PS 0-1
10. Willing to take biopsy before surgery and during chemotherapy and willing to take pre-operative chemotherapy and related treatment
11. Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to take an adequate contraceptive measure
12. Signed written informed consent; Able to comply with the protocol

Exclusion Criteria:

1. Prior systemic or loco-regional treatment of breast cancer, including chemotherapy
2. Metastatic breast cancer
3. Patients with medical conditions that renders them intolerant to neoadjuvant therapy and related treatment, including uncontrolled pulmonary disease, Diabetes Mellitus, severe infection, active peptic ulcer, Coagulation disorder, connective tissue disease or myelo-suppressive disease
4. History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (Systolic BP more than 180mmHg or Diastolic BP more than 100mmHg）
5. grade 1 peripheral neuropathy from any cause
6. Patient is pregnant or nursing
7. Not willing to take pre-operative biopsy or neo-adjuvant therapy
8. Patients with psychiatric disorder or other disease leading to incompliance to the therapy
9. Known hypersensitivity to any ingredient of the regimen
10. Treatment with any investigational drug within 30 days before the beginning of treatment with study drug

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint is efficacy. To compare the efficacy in terms of the pathological complete response rate (pCR) to preoperative administration of qw or q3w Paclitaxel, Carboplatin and Trastuzumab (PCH). | 3 years from last patient randomized
  Primary Endpoint is efficacy. To compare the efficacy in terms of the pathological complete response rate (pCR) to preoperative administration of qw or q3w Paclitaxel, Carboplatin and Trastuzumab (PCH). The primary efficacy variable is the rate of pathological complete response (pCR). Time to recurrence will be measured as the time from when the patient was randomized to the time the patient is first recorded as having disease recurrence or the date of death if the patient dies due to causes other than disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Post-Doctor, Principal Investigator — Cancer Hospital Affiliated to Fudan University
Locations (1):
- Cancer Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China